CLINICAL TRIAL: NCT05294172
Title: KL-A167 Injection Combined With Cisplatin and Gemcitabine vs Placebo Combined With Cisplatin and Gemcitabine in the Treatment of Recurrent or Metastatic Nasopharyngeal Carcinoma: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Clinical Trial
Brief Title: KL-A167 Injection Combined With Cisplatin and Gemcitabine vs Placebo Combined With Cisplatin and Gemcitabine in the Treatment of Recurrent or Metastatic Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KL-A167-III-08
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Nasopharyngeal Carcinoma; Recurrent or Metastatic
Keywords: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Recurrence; Neoplasm Metastasis | interventions — 18-O-demethylcervinomycin A2; Gemcitabine; Injections; Cisplatin

STUDY DESIGN:
Intervention Model Description: multicenter, double-blind, randomized, controlled phase III trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KL-A167+Gemcitabine+Cisplatin (Experimental): subject will receive KL-A167 1200mg every 3 weeks, cisplatin 80mg/m2 on Day 1 of each 21 day, 4-6 cycles, gemcitabine 1000mg/m2, Day 1 and Day 8 of each 21 day,4-6 cycles
  Interventions: Drug: KL-A167; Drug: Gemcitabine; Drug: Cisplatin
- Placebo+Gemcitabine+Cisplatin (Placebo Comparator): subject will receive placebo every 3 weeks, cisplatin 80mg/m2 on Day 1 of each 21 day, 4-6 cycles, gemcitabine 1000mg/m2, Day 1 and Day 8 of each 21 day, 4-6 cycles
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Placebo

INTERVENTIONS:
Drug: KL-A167 — KL-A167 4-6 cycles for combined therapy.KL-A167 maintenance.
  Arms: KL-A167+Gemcitabine+Cisplatin
Drug: Gemcitabine — 4-6 cycles for combined therapy
  Other Names: Gemcitabine Hydrochloride for Injection
Drug: Cisplatin — 4-6 cycles for combined therapy.
  Other Names: Cisplatin injection
Drug: Placebo — 4-6 cycles for combined therapy.Placebo maintenance.
  Arms: Placebo+Gemcitabine+Cisplatin

SUMMARY:
The study is to evaluate the efficacy of KL-A167 combined with cisplatin and gemcitabine vs placebo combined with cisplatin and gemcitabine in the treatment of recurrent or metastatic nasopharyngeal carcinoma, as measured by progression-free survival (PFS) per the Response Evaluation Criteria in Solid Tumors RECIST Version 1.1

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled and multicenter study. It is expected that patients with recurrent or metastatic nasopharyngeal carcinoma who had not received systematic anti-tumor treatment before are enrolled, and the efficacy and safety of KL-A167 injection combined with cisplatin and gemcitabine are compared with placebo combined with cisplatin and gemcitabine in the treatment of recurrent or metastatic nasopharyngeal carcinoma. Subjects who meet the enrollment requirements will be randomized to the trial group or the control group according to the ratio of 2:1. The stratification factors are: liver metastasis (with vs without) and ECOG score (0 vs 1)

ELIGIBILITY:
Inclusion Criteria:

* The ages at the time of signing the informed consent are ≥ 18 years old and ≤ 75 years old, regardless of gender.
* Patients with nasopharyngeal carcinoma diagnosed definitively by histology or cytology.
* Recurrent or metastatic nasopharyngeal carcinoma:Nasopharyngeal carcinoma patients with distant metastasis at the time of initial diagnosis (stage IVB nasopharyngeal carcinoma as defined by the 8th Edition of the staging system of Union for International Cancer Control and American Cancer Joint Committee); or nasopharyngeal carcinoma patients with local recurrence and/or distant metastasis more than 6 months after the end of previous radical treatment.Have not received systematic treatment for recurrent or metastatic nasopharyngeal carcinoma before; those who have local recurrence are not suitable for local treatment or have been treated locally.
* Eastern Cooperative Oncology Group (ECOG) performance status is 0 ~ 1 score, and the expected survival time is ≥ 12 weeks.
* At least one measurable lesion according to RECIST 1.1; the lesions that have received radiotherapy are not selected as target lesions.
* Patients must provide tissues or tissue specimens for biomarker analysis during the screening period, and the freshly obtained tissues are preferred. Patients who cannot obtain the fresh tissues can provide archived paraffin sections.
* Significant organ functions meet the following requirements:a)Blood routine: Neutrophil count (NEUT) ≥ 1.5×109/L; platelet count (PLT)≥100×109/L; hemoglobin ≥ 90 g/L.b)Liver function: Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal value (ULN); total bilirubin (TBIL) ≤ 1.5×ULN; for patients with liver metastasis, ALT and AST ≤ 5×ULN; for patients with liver metastasis or Gilbert syndrome, TBIL ≤ 3×ULN.c)Albumin ≥ 30 g/L.d)Renal function: creatinine clearance rate (CrCl) ≥ 60 ml/min (using standard Cockcroft-Gault formula).e)Coagulation function: International standardized ratio (INR) ≤ 1.5×ULN; activated partial thromboplastin time (APTT) ≤ 1.5×ULN.
* Those who have child-bearing potential during the study period and within 6 months after the end of the last dose study (both men and women) must take effective medical contraceptive measures.
* Patients voluntarily participate in this study, sign informed consent, and are able to comply with the visits and related procedures specified in the protocol.

Exclusion Criteria:

* Patients with pathologically diagnosed nasopharyngeal adenocarcinoma or sarcoma.
* Central nervous system metastasis is present at the time of screening.
* Uncontrollable tumor-related pain.
* Other malignant tumors before randomization (except those who have non-melanoma in situ skin cancer, superficial bladder cancer, cervical cancer in situ, breast cancer, localized prostate cancer, etc., which have been cured and not recurred within 3 years, and the investigator considers those who can be enrolled).
* It is known that there is a history of allergy to any ingredient of KL-A167 injection or severe hypersensitivity to other monoclonal antibodies, or hypersensitivity to gemcitabine, cisplatin and any excipients.
* Have received any of the following treatment:a)Previous immunotherapy, including immune checkpoint inhibitors (such as PD-1 antibody, PD-L1 antibody, CTLA-4 antibody, etc.), immune checkpoint agonists, immune cell therapy and other treatments targeting at the immune mechanism of tumor.b)Any clinical study drugs within 4 weeks before randomization.c)Participation in another clinical study concurrently, unless it is an observational (non-interventional) clinical study or an interventional clinical study follow-up.d)The last dose of non-systemic anticancer therapy (including local radiotherapy, radiofrequency ablation, anti-tumor Chinese patent medicine, etc.) within 2 weeks before randomization.e)Those who were vaccinated with anti-tumor vaccine previously or have been vaccinated with any active vaccine (such as influenza vaccine, varicella vaccine, etc.) within 4 weeks before randomization or plan to do so during the study period.f)Major surgery (except diagnosis of nasopharyngeal carcinoma) or severe trauma was performed within 4 weeks before randomization.g)Any blood components, anemia correcting drugs (including but not limited to drugs which supplement hematopoietic raw materials, raise red blood cells and raise hemoglobin), drugs which raise white blood cells and platelets were used within 2 weeks before randomization.
* Concomitant diseases that may affect protocol compliance or trial results, including:a)Major cardiovascular diseases, such as Grade II and above cardiac dysfunction (NYHA standard); myocardial infarction, unstable arrhythmia or unstable angina pectoris within 3 months before randomization; previous history of myocarditis or cardiomyopathy; echocardiography showed ejection fraction < 50%; QTc interval, male > 450 msec, female > 470 msec; ECG examination is abnormal and the investigator considers there is additional risk.b) Symptomatic hypercalcemia (serum calcium> 2.9 mmol/L ).
* The toxicity of previous anti-tumor treatment has not recovered to ≤ CTCAE version 5.0 Level 1 or the level specified in the inclusion/exclusion criteria (except for hair loss, fatigue, sequelae of neurotoxicity related to previous platinum treatment, specific laboratory investigation abnormalities and other conditions that the investigator judges there is no safety risk).
* The history of allogeneic organ transplantation or hematopoietic stem cell transplantation is known.
* Severe chronic or active infections (including active tuberculosis, etc.) occurred within 2 weeks before randomization, which required systemic antibiotics or antiviral treatment.
* Any patient with active autoimmune disease or a history of autoimmune disease and possible recurrence, including but not limited to neurological diseases related to immunity, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel diseases including Crohn's disease and ulcerative colitis, autoimmune hepatitis, toxic epidermal necrolysis (TEN) or Stevens-Johnson syndrome.Note: Patients with the following diseases are not excluded, and can be screened following other inclusion and exclusion criteria:a)Type 1 diabetes that can be controlled by stable dose of insulin.b)Hypothyroidism that can be controlled by hormone replacement therapy alone.c)Skin diseases that do not require systemic treatment (e.g. vitiligo, psoriasis, hair loss).d)Any other disease that is not expected to recur in the absence of external triggers.
* Treated with systemic immuno-agonists (including but not limited to interferon or IL-2) or received systemic treatment with steroid hormones (equivalent to prednisone > 10 mg/day) or other immunosuppressants within 2 weeks before randomization.Note: Subjects without active immune diseases are allowed to receive steroid hormone replacement therapy with a dose equivalent to prednisone ≤ 10 mg/day. Topical, intraocular, intra-articular, intranasal or inhaled corticosteroids (extremely low systemic absorption) are allowed; short-term use of corticosteroids is allowed to prevent (such as allergy to contrast media) or treat non-autoimmune conditions (such as delayed type hypersensitivity caused by exposure to allergens).
* Patients have active hepatitis B (HBsAg positive, but if HBV DNA detected by each study site ≤ 1×103 copy number/ml or lower than the lower limit of reference value, patients are allowed to be enrolled) or hepatitis C (hepatitis C antibody positive, but if HCV RNA lower than the lower limit of detection method, patients are allowed to be enrolled).
* The history of positive test for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) is known.
* For patients with known history of interstitial lung disease (such as idiopathic pulmonary fibrosis, sarcoidosis, etc.) and non-infectious pneumonia (such as intensified pneumonia, idiopathic pneumonia, etc.), those who had drug-induced or radiation-induced rather than infectious pneumonia but were asymptomatic are allowed to be enrolled in the group.
* Grade 2 or above peripheral nerve disease , defined according to CTCAE 5.0 standard.
* Pregnant or lactating women.
* Other clinically significant underlying diseases that may affect drug administration and protocol compliance (such as poorly controlled diabetes/hypertension, pleural effusion/pericardial effusion/ascites requiring repeated drainage, drug or alcohol abuse, etc.) considered by the investigator, as well as other factors that may affect the efficacy or safety assessment of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 24 month
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the Independent Review Committee according to RECIST v1.1 or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Progression-free survival(PFS) | up to 24 month
  Progression-free survival (PFS) assessed by the investigators according to RECIST V 1.1
Objective Response Rate (ORR) | up to 24 month
  The percentage of patients with CR and PR assessed by the Independent Review Committee and investigators according to RECIST v 1.1
Disease Control Rate (DCR) | up to 24 month
  The proportion of patients who have achieved CR，PR and SD assessed by the Independent Review Committee and investigators according to RECIST v 1.1
Duration of Response (DoR) | up to 24 month
  From the date that response criteria are first met to the first occurrence of PD as determined by the Independent Review Committee and investigators according to RECIST v1.1 or death from any cause, whichever occurs first
Overall Survival (OS) | up to 24 month
  OS, defined as the time from randomization to death or lose of follow, whichever occurs first
1 year and 2 years Overall Survival (OS) rate | up to 24 month
  The percentage of patients overall survival in 1 year and 2 years
Time to Response（TTR） | up to 24 month
  The time from randomization to the date that response criteria are first met assessed by the Independent Review Committee and investigators according to RECIST v 1.1

OTHER OUTCOMES:
Progression-free survival(PFS) | up to 24 month
  PFS, defined as the active comparator arm frist dosing of KL-A167 injection to the first occurrence of disease progression as determined by the investigators according to RECIST v1.1 or death from any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No